CLINICAL TRIAL: NCT01648075
Title: Effect of the Consumption of Probiotics Lactobacilli Enriched Milk in the Reduction of Incidence of Carious Lesions in Preschool Children
Brief Title: Effect of the Consumption of Probiotics in the Reduction of Incidence of Carious Lesions in Preschool Children
Acronym: Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Gonzalo Rodriguez, DDS, Effect of the consumption of probiotics lactobacilli enriched milk in the reduction of incidence of carious lesions in preschool children, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Universidad de Chile
Record Dates: First submitted 2012-07-09; First posted 2012-07-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Caries Reduction; Caries Prevention
Keywords: caries; probiotics; lactobacilli

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Probiotic enriched milk (Experimental): 150 ml of skimmed milk enriched with probiotic (Lactobacillus rhamnosus LRH08) once a day
  Interventions: Dietary Supplement: Experimental: Probiotic enriched milk
- Skimmed Milk (Placebo Comparator): 150 ml of skimmed milk once a day
  Interventions: Dietary Supplement: Experimental: Probiotic enriched milk

INTERVENTIONS:
Dietary Supplement: Experimental: Probiotic enriched milk — Milk will be enriched with lactobacillus rhamnosus for the experimental group.
  Other Names: probiotic: Lactobacillus rhamnosus

SUMMARY:
Probiotics are microorganisms that when administered in adequate amounts can confer health benefits. In vitro and clinical studies support the idea that lactobacilli have protective effects on oral health. A recent study in which preschoolers consumed milk drinks enriched with Lactobacillus rhamnosus, reported a reduction in caries, as well as additional benefits to children.

The aim of this study is to evaluate the effect of daily consumption of milk beverages enriched with Lactobacillus rhamnosus on the incidence of caries in preschool Chilean children.

DETAILED DESCRIPTION:
In this randomized controlled trial, preschool children belonging to Integra Foundation will be invited to participate. After obtaining parent´s informed consent, clinical and microbiological testing of saliva at baseline, 6 m, 12m and 18m will be performed. Differences in prevalence and incidence of caries, dmft and microbial diversity between groups will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children from a general health perspective, with or without cavitated carious lesions at baseline.

Exclusion Criteria:

* Children with systemic disorders who need special care and / or who have intolerance to milk drinks or allergy to any of the components of the experimental and / or placebo beverage.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Reduction of caries incidence in 1 unit of DMF-T (decayed, missing and filled teeth) from baseline up to the 18th month | 18 months
  Preschool children that in regular basis consume enriched milk with probiotics will present less caries incidence than those that consume milk without probiotics, measured by differences in dmft index between baseline, 6 months, 12 months and 18 months dental exams.

CONTACTS AND LOCATIONS:
Locations (1):
- Integra Preschools, Santiago, Metropolitan Region, Chile

REFERENCES:
- [Derived] Ibacache RC, Faleiros S, Diaz-Dosque M, Ruiz B, Contador R, Moreno B, Godoy EF, Martinez GR. Effect of probiotic supplementation on the progression of non-cavitated carious lesions in children: A 12-month randomized controlled trial. Eur J Oral Sci. 2025 Dec 15:e70061. doi: 10.1111/eos.70061. Online ahead of print. PMID 41398922
- [Derived] Rodriguez G, Ruiz B, Faleiros S, Vistoso A, Marro ML, Sanchez J, Urzua I, Cabello R. Probiotic Compared with Standard Milk for High-caries Children: A Cluster Randomized Trial. J Dent Res. 2016 Apr;95(4):402-7. doi: 10.1177/0022034515623935. Epub 2016 Jan 8. PMID 26747421